CLINICAL TRIAL: NCT03904147
Title: Clinical Trial to Evaluate Cardiovascular Outcomes In Patients Treated With the Tricuspid Valve Repair System Pivotal
Brief Title: TRILUMINATE Pivotal Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-CIP-10249
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Tricuspid Regurgitation
Keywords: ABT-CIP-10249; Tricuspid; Cardiovascular; Pivotal
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Randomized - Device Group (Experimental): Subjects will undergo TriClip implantation and will continue to be managed on medical therapy, per physician discretion
  Interventions: Device: TriClipTM Device
- Randomized - Control Group (Active Comparator): Subjects will continue to be managed on medical therapy, per physician discretion
  Interventions: Device: TriClipTM Device
- Single Arm Group (Experimental): Subjects will receive the TriClip device and will continue to be managed on medical therapy, per physician discretion.
  Interventions: Device: TriClipTM Device
- Continued Access Study (CAS) (Experimental): Subjects will undergo TriClip implantation and will continue to be managed on medical therapy, per physician discretion
  Interventions: Device: TriClipTM Device

INTERVENTIONS:
Device: TriClipTM Device — Transcatheter TriClip placement in the tricuspid valve to repair the valve and correct regurgitation

SUMMARY:
The primary objective of this trial is to demonstrate the safety and effectiveness of the TriClip device in improving clinical outcomes in symptomatic patients with severe tricuspid regurgitation (TR), who are at intermediate or greater estimated risk for mortality or morbidity with tricuspid valve surgery. This randomized controlled trial will compare the investigational device (TriClip device) to Control (Medical Therapy).

ELIGIBILITY:
Inclusion Criteria:

* In the judgment of the site local heart team, subject has been adequately treated per applicable standards (including medical management) and stable for at least 30 days as follows:

  * Optimized medical therapy for treatment of TR (e.g. diuretics).
  * Medical and/or device therapy, for mitral regurgitation, atrial fibrillation, coronary artery disease and heart failure.
  * The Eligibility Committee will confirm that the subject has been adequately treated medically.
* Subject is symptomatic with Severe TR despite being optimally treated as described above. TR severity is determined by the assessment of a qualifying TTE and confirmed by the ECL. The ECL will also request a TEE to confirm TR etiology. Note: If any cardiac procedure(s) occur after eligibility was determined, TR severity will need to be re-assessed 30 days after the cardiac procedure(s).
* The cardiac surgeon of the site local heart team concur that the patient is at intermediate or greater estimated risk for mortality or morbidity with tricuspid valve surgery.
* New York Heart Association (NYHA) Functional Class II, III or ambulatory class IV
* In the judgment of the TriClip(TM) implanting Investigator, femoral vein access is determined to be feasible and can accommodate a 25 Fr catheter.
* Age ≥18 years at time of consent.
* Subject must provide written informed consent prior to any trial related procedure.

Exclusion Criteria:

* Systolic pulmonary artery pressure (sPAP) > 70 mmHg or fixed pre-capillary pulmonary hypertension as assessed by right heart catheterization (RHC)
* Severe uncontrolled hypertension Systolic Blood Pressure (SBP) ≥ 180 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 110 mm Hg
* Any prior tricuspid valve procedure that would interfere with placement of the TriClip(TM) device
* Indication for left-sided (e.g. severe aortic stenosis, severe mitral regurgitation) or pulmonary valve correction prior 60 days. Note: Patients with concomitant Mitral and tricuspid valve disease will have the option of getting their MR treated, and wait 60 days prior to being reassessed for the trial.
* Pacemaker or ICD leads that would prevent appropriate placement of the TriClip(TM) clip.
* Tricuspid valve stenosis - Defined as a tricuspid valve orifice of ≤ 1.0 cm2 and/or mean gradient ≥5 mmHg as measured by the ECL
* Left Ventricular Ejection Fraction (LVEF) ≤20%
* Tricuspid valve leaflet anatomy which may preclude clip implantation, proper clip positioning on the leaflets or sufficient reduction in TR. This may include:

  * Evidence of calcification in the grasping area
  * Presence of a severe coaptation defect (> 2cm) of the tricuspid leaflets
  * Severe leaflet defect(s) preventing proper device placement
  * Ebstein Anomaly - Identified by having a normal annulus position while the valve leaflets are attached to the walls and septum of the right ventricle.
* Tricuspid valve anatomy not evaluable by TTE and TEE
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e. noncompliant, perforated).
* MI or known unstable angina within prior 30 days
* Percutaneous coronary intervention within prior 30 days
* Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
* Cerebrovascular Accident (CVA) within prior 90 days
* Chronic dialysis
* Bleeding disorders or hypercoagulable state
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Contraindication, allergy or hypersensitivity to dual antiplatelet and anticoagulant therapy.

  * Note: Contraindication to either antiplatelet or anticoagulant therapy (individually not both therapies) is not an exclusion criterion.
* Ongoing infection requiring current antibiotic therapy (if temporary illness, patients may enroll 30 days after discontinuation of antibiotics with no active infection).
* Known allergy or hypersensitivity to device materials
* Evidence of intracardiac, inferior vena cava (IVC), or femoral venous mass, thrombus or vegetation.
* Life expectancy of less than 12 months
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
* Subject is currently participating in another clinical investigation for valvular heart disease(s).
* Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period. Female subjects of child-bearing potential are required to have a negative pregnancy test done within 7 days of the baseline visit per site standard test. Female patients of childbearing potential should be instructed to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release.) It is accepted, in certain cases, to include subjects having a sterilized regular partner or subjects using a double barrier contraceptive method.
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2029-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Griffin, PhD, Study Director — Abbott Structural Heart; David Adams, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Paul Sorajja, MD, Principal Investigator — Allina Health System
Locations (76):
- United States (63):
  - University Hospital - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Scripps Green Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Providence Medical Foundation (St. Joseph Hospital), Orange, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - University of California - Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven, New Haven, Connecticut
  - JFK Medical Center, Atlantis, Florida
  - Manatee Memorial Hospital, Bradenton, Florida
  - Morton Plant Valve Clinic, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Palm Beach Garden Medical Center, Palm Beach Gardens, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Albany Medical Center, Albany, New York
  - Buffalo General Hospital, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - Methodist Hospital of San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin
- Canada (7):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Science Centre, Hamilton, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - The Royal Victoria, Montreal, Quebec
- Germany (4):
  - München Grosshadern, München, Bavaria
  - Universitätsklinikum Bonn AdöR, Bonn, North Rhine-Westphalia
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
- Ospedale San Raffaele - Cardiac, Milan, Lombard, Italy
- Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kar S, Makkar RR, Whisenant BK, Hamid N, Naik H, Tadros P, Price MJ, Singh G, Schwartz JG, Kapadia S, Alli O, Horr S, Seshiah P, Batchelor W, Jones BM, Ahmed MI, Benza R, Jorde U, Thourani VH, Ghobrial AA, Tang GHL, Trusty PM, Huang D, Hahn RT, Adams DH, Sorajja P; TRILUMINATE Pivotal Investigators. Two-Year Outcomes of Transcatheter Edge-to-Edge Repair for Severe Tricuspid Regurgitation: The TRILUMINATE Pivotal Randomized Controlled Trial. Circulation. 2025 Jun 10;151(23):1630-1638. doi: 10.1161/CIRCULATIONAHA.125.074536. Epub 2025 Mar 30. PMID 40159089
- [Derived] Naik H, Price MJ, Kapadia S, Whisenant BK, Tadros P, Makkar R, Asgar AW, Fam N, Tang GHL, Mehta SR, Byrne T, Singh G, Panaich SS, Peterman K, Trusty PM, Hamid N, Hahn RT, Adams DH, Sorajja P. Tricuspid Transcatheter Edge-to-Edge Repair in Patients With Transvalvular CIED Leads: The TRILUMINATE Pivotal Trial. JACC Clin Electrophysiol. 2025 May;11(5):1012-1020. doi: 10.1016/j.jacep.2025.01.001. Epub 2025 Jan 20. PMID 39903153
- [Derived] Cavalcante JL, Scherer M, Fukui M, Lerakis S, Harb S, Pursnani A, Schwartz JG, Kapadia S, Ricciardi MJ, Khalique O, Kodali S, Shah D, Little SH, Sekaran N, Whisenant B, Flueckiger P, Yadav P, Emaminia A, Batchelor W, Kellman P, Lin Z, Trusty PM, Hahn RT, Adams D, Sorajja P. Advanced Imaging Assessment of the Impact of Tricuspid Regurgitation on Cardiac Remodeling: The TRILUMINATE Pivotal Imaging Substudy. J Am Coll Cardiol. 2025 Jan 28;85(3):250-261. doi: 10.1016/j.jacc.2024.09.009. Epub 2024 Nov 20. PMID 39570246
- [Derived] Jorde UP, Benza R, McCarthy PM, Ailawadi G, Whisenant B, Makkar R, Tadros P, Naik H, Fam N, Sauer AJ, Murthy S, Kar S, von Bardeleben RS, Hahn RT, Hamid N, Zbinden J, Sorajja P, Adams D. Impact of Renal and Liver Function on Clinical Outcomes Following Tricuspid Valve Transcatheter Edge-to-Edge Repair. J Am Coll Cardiol. 2024 Dec 17;84(25):2446-2456. doi: 10.1016/j.jacc.2024.08.044. Epub 2024 Aug 31. PMID 39222896
- [Derived] Sorajja P, Whisenant B, Hamid N, Naik H, Makkar R, Tadros P, Price MJ, Singh G, Fam N, Kar S, Schwartz JG, Mehta S, Bae R, Sekaran N, Warner T, Makar M, Zorn G, Spinner EM, Trusty PM, Benza R, Jorde U, McCarthy P, Thourani V, Tang GHL, Hahn RT, Adams DH; TRILUMINATE Pivotal Investigators. Transcatheter Repair for Patients with Tricuspid Regurgitation. N Engl J Med. 2023 May 18;388(20):1833-1842. doi: 10.1056/NEJMoa2300525. Epub 2023 Mar 4. PMID 36876753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The last 12-month follow-up visit for the 350 randomized subjects (primary analysis cohort) occurred on November 18, 2022. The last 12-month follow-up visit for the 100 Single-arm subjects (primary analysis cohort) occurred on November 1, 2022. Follow-up through 5years is ongoing for all cohorts.
Groups:
- Randomized - Device Group: Subjects will undergo TriClipTM implantation and will continue to be managed on medical therapy, per physician discretion
- Single Arm Group: Subjects will receive the TriClip TM device and will continue to be managed on medical therapy, per physician discretion.
Period: Overall Study
Arm/Group | Randomized - Device Group | Randomized - Control Group | Single Arm Group
Started | 175 | 175 | 100
Completed | 152 | 149 | 84
Not Completed | 23 | 26 | 16
Not completed — Death | 15 | 13 | 15
Not completed — Withdrawal by Subject | 7 | 12 | 1
Not completed — 1Y visit completed after 365 days | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized - Device Group | Randomized - Control Group | Single Arm Group | Total
Number analyzed (Participants) | 175 | 175 | 100 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (7.4) | 77.8 (7.2) | 80.4 (6.2) | 78.5 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 94 | 53 | 245
  Male | 77 | 81 | 47 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 4 | 18
  Not Hispanic or Latino | 163 | 153 | 94 | 410
  Unknown or Not Reported | 7 | 13 | 2 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 7 | 7 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 10 | 7 | 24
  White | 149 | 143 | 87 | 379
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 15 | 3 | 29
Prior Aortic or Mitral Valve Intervention [Count of Participants; unit: Participants] | 68 | 61 | 44 | 173

OUTCOME MEASURES:

1. Primary Outcome: For Randomized Cohort: Hierarchical Composite of All-cause Death or Tricuspid Valve Surgery, Heart Failure Hospitalizations, and KCCQ Improvement
Description: Analysis of hierarchical composite of all-cause death or tricuspid valve surgery, heart failure hospitalizations, and KCCQ improvement of at least 15 points was performed in ITT population using Finkelstein-Schoenfeld method.
  A win ratio was also calculated to descriptively quantify the magnitude of treatment benefits. The win ratio is calculated as the ratio of the number of wins in Device versus Control patients. The primary analysis population consisted of 175 Device patients and 175 Control patients, resulting in 30,625 Device-Control patient pairs (i.e., 175 × 175).
Time Frame: 12 Months
Measure: Number; unit: wins in the patient pairs
Groups:
- Randomized - Device Group: Subjects received Device treatment.
- Randomized - Control Group: Subjects received medical therapy alone.
Arm/Group | Randomized - Device Group | Randomized - Control Group
Number analyzed (Participants) | 175 | 175
wins in the patient pairs | 11,246 | 7,791
Statistical Analysis 1: Comparison: Randomized - Device Group vs Randomized - Control Group; Test type: Superiority; p = 0.0311, Finkelstein-Schoenfeld Method; Win Ratio = 1.44 — The Win Ratio provides an estimation of the treatment effect

2. Primary Outcome: For Single-Arm Cohort: Rate of Survival Through 12 Months With a Quality of Life Improvement (Assessed Using KCCQ Overall Score) of at Least 10 Points Compared to Baseline.
Description: This outcome will be assessed as the percentage of subjects meeting the definition of the endpoint.
Time Frame: 12 months
Population: Nine (9) subjects were not included in the primary endpoint analysis due to:
  * KCCQ not available at 12-month visit (n=6)
    * Subject missed 12-month visit (n=3)
    * Subject declined to complete KCCQ (n=2)
    * Subject did not complete a 12-month visit due to COVID-19 (n=1)
  * Subject experienced hospitalization or death related to COVID-19 prior to 12-month follow-up visit (n=2)
  * Subject withdrew prior to 12-month visit (n=1)
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Group
Number analyzed (Participants) | 91
percentage of participants | 46.2
Statistical Analysis 1: Comparison: Single Arm Group; Test type: Superiority; p = 0.0008, exact test

3. Secondary Outcome: For Randomized Cohort - Device Group Only: Rate of Kaplan-Meier Estimate (SE) of Freedom From Major Adverse Events (MAE) Occurring Within 30 Days Post-procedure
Description: Freedom from major adverse events (MAE) was assessed in the Attempted Procedure population (n=172). MAEs included cardiovascular mortality, new onset renal failure, endocarditis requiring surgery, and non-elective cardiovascular surgery for TriClip device-related AE post-index procedure.
Time Frame: 30 Days
Measure: Number; unit: percentage of participants
Arm/Group | Randomized - Device Group
Number analyzed (Participants) | 172
percentage of participants | 98.3
Statistical Analysis 1: Comparison: Randomized - Device Group; Test type: Superiority; p < 0.0001, Z test

4. Secondary Outcome: For Randomized Cohort: Change in Quality of Life as Assessed by KCCQ Score
Description: The mean change in KCCQ score between 12 months and baseline in the Device and Control groups will be compared, while adjusting for the baseline KCCQ score. The primary analysis for this endpoint imputed a KCCQ score of 0 at 12-month visit for all subjects who experienced a heart failure related cardiovascular death or received tricuspid valve surgery prior to completing 12-month follow-up. All KCCQ scores are scaled from 0 (worst) to 100 (best possible status), where the higher score reflects a better health status.
Time Frame: 12 months minus baseline
Population: Forty (11%) of the 350 subjects (20 Device, 20 Control) were not included in this endpoint due to missing paired KCCQ values at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Randomized - Device Group | Randomized - Control Group
Number analyzed (Participants) | 155 | 155
scores on a scale | 12.0 (25.8) | 1.0 (21.0)
Statistical Analysis 1: Comparison: Randomized - Device Group vs Randomized - Control Group; Test type: Superiority; p < 0.0001, ANCOVA model

5. Secondary Outcome: For Randomized Cohort: Tricuspid Regurgitation Reduction to Moderate or Less at 30-Day Visit
Description: The percentage of subjects with tricuspid regurgitation reduced to moderate or less at 30-day visit in the Device Group will be compared with that in the Control Group. Tricuspid regurgitation severity will be graded on a 5-point scale: trace/mild, moderate, severe (severe 3), massive (severe 4), and torrential (severe 5), which has frequently been used in recent interventional tricuspid studies to categorize tricuspid regurgitation severity. This grading system follows the 2017 ASE guidelines (Zoghbi WA, Adams D, Bonow RO et al. Recommendations for Noninvasive Evaluation of Native Valvular Regurgitation: A Report from the American Society of Echocardiography Developed in Collaboration with the Society for Cardiovascular Magnetic Resonance. J Am Soc Echocardiogr 2017;30:303-371.), and further stratifies the traditional "severe" category into severe (Severe 3), massive (Severe 4), and torrential (Severe 5).
Time Frame: 30 Days
Population: Forty-one (41, or 12%) of the 350 subjects (13 Device, 28 Control) were not included in the analysis of this endpoint due to TR not available at 30 days.
Measure: Number; unit: percentage of participants
Groups:
- Randomized -Control Group: Subjects will continue to be managed on medical therapy, per physician discretion
Arm/Group | Randomized - Device Group | Randomized -Control Group
Number analyzed (Participants) | 162 | 147
percentage of participants
  Trace | 10.5 | 0.7
  Mild | 39.5 | 0.7
  Moderate | 37.0 | 4.1
  Severe 3 | 11.1 | 22.4
  Severe 4 | 0.6 | 21.8
  Severe 5 | 1.2 | 50.3
Statistical Analysis 1: Comparison: Randomized - Device Group vs Randomized -Control Group; Test type: Superiority; p < 0.0001, Chi-square test

6. Secondary Outcome: For Randomized Cohort: Change in 6 Minute Walk Test (6MWT) From Baseline to 12 Months
Description: The primary analysis for this endpoint imputed a 6MWT distance of 0 meters for all subjects who experienced a heart failure related cardiovascular death or received tricuspid valve surgery prior to completing 12-month follow-up. Subjects who were unable to exercise due to cardiac reasons were also assigned a 6MWT distance of 0 meters at 12-month follow-up. Other subjects with missing 6MWT distance at either baseline or 12-month follow-up were excluded from the analysis.
Time Frame: 12 Months
Population: Eighty-three (24%) of the 350 subjects (44 Device, 39 Control) were not included in this endpoint due to missing paired 6MWT values at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Randomized - Device Group | Randomized - Control Group
Number analyzed (Participants) | 131 | 136
meters | -5.1 (131.4) | -28.1 (122.3)
Statistical Analysis 1: Comparison: Randomized - Device Group vs Randomized - Control Group; Test type: Superiority; p = 0.2482, ANCOVA model

7. Secondary Outcome: For Single-Arm Cohort: The Percentage of Subjects With TR Reduction by at Least 1 Grade at 30-Day Follow-up
Time Frame: 30 days
Population: Twelve subjects were not included in the analysis of this endpoint due to missing paired TR severity at baseline and 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Group
Number analyzed (Participants) | 88
percentage of participants | 98.9
Statistical Analysis 1: Comparison: Single Arm Group; Test type: Superiority; p < 0.0001, Exact test

8. Secondary Outcome: For Single-Arm Cohort: Rate of Freedom From MAE Through 30 Days
Description: Freedom from MAE occurring after procedure attempt (femoral vein puncture) at 30 days. Components of MAE consist of Cardiovascular Mortality, New Onset Renal Failure, Endocarditis Requiring Surgery, and Non-Elective Cardiovascular Surgery for TriClip device-related AE post-index procedure.
Time Frame: 30 days
Population: One subject (Subject 1300) withdrew from the study prior to 30 days without experiencing any MAE and was therefore excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Group
Number analyzed (Participants) | 99
percentage of participants | 100.0
Statistical Analysis 1: Comparison: Single Arm Group; Test type: Superiority; p < 0.0001, Binomial exact method

9. Secondary Outcome: For Single-Arm Cohort: Change in 6 Minute Walk Test (6MWT) From Baseline to 12 Months
Description: This analysis imputed a 6MWT distance of 0 meters for all subjects who were unable to exercise due to cardiac reasons. However, there were no subjects unable to exercise due to cardiac reasons and therefore no imputation was performed. Subjects with missing 6MWT distance at either baseline or 12-month follow-up were excluded from the analysis.
Time Frame: 12 months
Population: Twenty-nine (29%) subjects were not included in the primary analysis due to missing 6MWT values at baseline and/or 12 months.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Single Arm Group
Number analyzed (Participants) | 71
meter | 13.7 (92.7)
Statistical Analysis 1: Comparison: Single Arm Group; Test type: Superiority; p = 0.1090, normal approximation

10. Secondary Outcome: Recurrent HF Hospitalizations at 24 Months
Description: H0: HR(24M)>1; H1: HR(24M)≤1
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2024-12

11. Secondary Outcome: Freedom From All-cause Mortality, Tricuspid Valve Surgery, and Tricuspid Valve Intervention at 24 Months
Description: H0: Survival curves of the two groups through 24 months are the same. H1: Survival curves of the two groups through 24 months are different.
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 12 months
Description: The participant flow reports patient status based on visit windows in order to report if a patient completed a visit or not. The AE section including the All-Cause Mortality reports all events through 365 days.
Groups:
- Randomized - Single Arm Group: Subjects will receive the TriClip TM device and will continue to be managed on medical therapy, per physician discretion.
Arm/Group | Randomized - Device Group | Randomized - Control Group | Randomized - Single Arm Group
All-Cause Mortality (participants affected / at risk) | 15/175 | 13/175 | 15/100
Serious Adverse Events (participants affected / at risk) | 85/175 | 73/175 | 62/100
Other Adverse Events (participants affected / at risk) | 29/175 | 28/175 | 33/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized - Device Group (N=175) | Randomized - Control Group (N=175) | Randomized - Single Arm Group (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 3 | 6
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 0 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 10 | 7 | 4
ATRIAL FLUTTER (Cardiac disorders) | 1 | 2 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 3 | 1 | 2
CARDIAC ARREST (Cardiac disorders) | 0 | 2 | 1
CARDIAC FAILURE (Cardiac disorders) | 26 | 20 | 21
CARDIAC FAILURE ACUTE (Cardiac disorders) | 2 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 0 | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 2
CHORDAE TENDINAE RUPTURE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 2 | 1 | 1
SINUS ARREST (Cardiac disorders) | 1 | 0 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 6 | 7 | 11
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
ADRENAL MASS (Endocrine disorders) | 1 | 0 | 0
HYPOPARATHYROIDISM (Endocrine disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 3 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 2 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
TONGUE HAEMATOMA (Gastrointestinal disorders) | 0 | 0 | 1
ASTHENIA (General disorders) | 2 | 0 | 2
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 1 | 1 | 0
DEATH (General disorders) | 2 | 3 | 2
DEVICE DEPLOYMENT ISSUE (General disorders) | 3 | 1 | 1
MULTI-ORGAN FAILURE (General disorders) | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 1
OTHERS (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 1 | 1
THROMBOSIS IN RIGHT ATRIAL LEAD (General disorders) | 1 | 0 | 0
CHOLANGITIS (Hepatobiliary disorders) | 0 | 0 | 1
AMYLOIDOSIS (Immune system disorders) | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 4 | 3
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 2
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
INFECTION (Infections and infestations) | 0 | 0 | 2
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
MENINGOENCEPHALITIS HERPETIC (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 1 | 2
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 | 0 | 0
PULMONARY SEPSIS (Infections and infestations) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 4 | 2 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 2 | 2
UROSEPSIS (Infections and infestations) | 0 | 1 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 5 | 3
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 0
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0 | 0
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0
CATHETERISATION CARDIAC (Investigations) | 0 | 1 | 0
CORONAVIRUS TEST POSITIVE (Investigations) | 1 | 0 | 1
ECHOCARDIOGRAM ABNORMAL (Investigations) | 0 | 1 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 1
TROPONIN INCREASED (Investigations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 1 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INGUINAL MASS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 | 2 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 2 | 0
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 | 0 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 1 | 0
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 1 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1 | 0
SYNCOPE (Nervous system disorders) | 4 | 0 | 0
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 0 | 2
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0
NEPHROPATHY (Renal and urinary disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 7 | 5 | 9
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
EXERCISE LACK OF (Social circumstances) | 0 | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 | 0 | 1
MEDICAL DEVICE IMPLANTATION (Surgical and medical procedures) | 0 | 1 | 0
ROTATOR CUFF REPAIR (Surgical and medical procedures) | 0 | 0 | 1
STENT PLACEMENT (Surgical and medical procedures) | 0 | 0 | 1
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 1 | 0 | 0
TRICUSPID VALVE REPAIR (Surgical and medical procedures) | 1 | 0 | 0
AORTIC STENOSIS (Vascular disorders) | 0 | 1 | 0
HAEMORRHAGE (Vascular disorders) | 14 | 7 | 8
HYPERTENSION (Vascular disorders) | 2 | 0 | 0
HYPOTENSION (Vascular disorders) | 5 | 0 | 4
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 1 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 0 | 1
SHOCK (Vascular disorders) | 0 | 0 | 1
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized - Device Group (N=175) | Randomized - Control Group (N=175) | Randomized - Single Arm Group (N=100)
ATRIAL FIBRILLATION (Cardiac disorders) | 5 | 1 | 5
CARDIAC FAILURE (Cardiac disorders) | 6 | 9 | 9
RENAL FAILURE ACUTE (Renal and urinary disorders) | 6 | 3 | 10
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 4
HAEMORRHAGE (Vascular disorders) | 9 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03904147/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03904147/SAP_001.pdf